CLINICAL TRIAL: NCT04453592
Title: The Effect of an Adductor Longus Tenotomy on the Bent Knee Fall Out Test
Brief Title: Adductor Longus Tenotomy & the BKFO Test
Status: Completed | Type: Observational
Sponsor: Aspetar (Other)
Collaborators: Clinique du sport (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALTBKFO
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Adductor Tendinitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention assigned as part of this study. — The intervention included in this study is part of routine medical care, and not assigned as a result of study participation. This study includes only the addition of a measurement; the bent knee fall out test. Therefore, we believe this study design is observational, and in line with the provided observation study design definition: "Observational: studies in human beings in which biomedical and/or health outcomes are assessed in predefined groups of individuals. Participants in the study may receive diagnostic, therapeutic, or other interventions, but the investigator does not assign specific interventions to the study participants. This includes when participants receive interventions as part of routine medical care, and a researcher studies the effect of the intervention."
  See uploaded study protocol for further details.

SUMMARY:
The bent knee fall out test (BKFO) is a common test for hip adductor flexibility. It is unknown whether the BKFO actually tests the the adductors or potentially hip range of motion instead.

In this study, the BKFO test is performed in the operating theater before and after an adductor longus tenotomy.

DETAILED DESCRIPTION:
Adductor-related groin pain is the most common type of groin pain in athletes, and pain at the proximal adductor longus insertion is a key finding in the diagnosis of longstanding groin pain. "Tightness" or "shortening" of the adductor longus is considered both a cause and effect of pain, that can lead to increased tension at the proximal insertion, thus playing a role in the persistence of longstanding adductor-related pain. For patients who do not respond sufficiently to non-surgical procedures, an adductor longus tenotomy is a surgical option that is considered to reduce tension at the proximal adductor longus insertion assisting in reduction of pain and return to sport.

The bent knee fall out test (BKFO) is one of the most commonly used tests to test adductor flexibility. This test involves a combined hip movement with hip flexion, abduction, and external rotation, and a high result is generally considered to be related to adductor muscle "tightness", specifically that of the adductor longus. It is uncertain whether the BKFO test is actually measuring adductor muscle flexibility or hip joint range of motion, as the test results may also be affected by a femoral head cam morphology. A slightly different test, called the Patrick FABER's test, involves a similar movement and is mainly used as a hip joint pain provocation test.

By cutting the adductor longus tendon, thereby removing the effect of potential adductor longus "tightness", it will be possible to show if and how much the flexibility of this muscle affects the BKFO test results. This will assist in future considerations of what this test is actually testing.

The aim of this study is to investigate the immediate effect of an adductor longus tenotomy on the results of the bent knee fall out test.

ELIGIBILITY:
Inclusion Criteria:

* adults (>18 years old)
* athletes (recreational or elite)
* clinical diagnosis of adductor-related groin pain
* patients undergoing unilateral or bilateral adductor longus tenotomy by one general surgeon.

Exclusion Criteria:

* No specific exclusion criteria were present other than refusal to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Athletes with groin pain are consecutively recruited from two clinics of a visceral surgeon specialized in groin pain in athletes. The clinics are located in Bordeaux and Paris, France, and patient population includes athletes from all over France.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du sport Bordeaux - Mérignac, Mérignac, France

IPD SHARING:
Plan to Share IPD: Undecided
There are currently no IPD plans. IPD data be obtained upon reasonable request

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenotomy: We included 60 male athletes consecutively between November 2019 and May 2020 all receiving an adductor longus tenotomy
Period: Overall Study
Arm/Group | Tenotomy
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Demographic Data of All Athletes: Demographic data (age, height, weight, BMI) for all included patients described in the baselines measures.
Arm/Group | Demographic Data of All Athletes
Number analyzed (Participants) | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age
  years | 27 [23 to 34.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 180.4 (7.8) [163 to 202]
Weight [Median (Inter-Quartile Range); unit: Kg] | 78 [71.5 to 85]
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 23.8 [22.2 to 26.2]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Bent Knee Fall Out Test
Description: The patient lies supine on the surgical table with app. 90° knee flexion, 45° hip flexion, and the feet together and the hips in external rotation (also known as the frog-leg position. Standardization of position is achieved by flexing one leg first, so the medial malleolus is placed next to the medial knee joint line of the contra-lateral leg. The knee is then moved laterally, externally rotating the hip with the plantar surface placed towards the contra-lateral leg. The contra-lateral leg is then flexed, and the plantar surfaces of the feet are aligned. The distance between the most distal point on the head of the fibula and the surface of the surgical table is measured using a rigid tape measure and distance is recorded in cm to the nearest 0.5 cm
Time Frame: Baseline pre-surgery and immediately after the surgery.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Tenotomy: all included patients
Arm/Group | Tenotomy
Number analyzed (Participants) | 60
cm | 3.9 (2)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events to report
Groups:
- Tenotomy: No adverse events in any patient
Arm/Group | Tenotomy
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT04453592/Prot_SAP_000.pdf